CLINICAL TRIAL: NCT07141966
Title: Assessment of Physical Activity, Balance, Muscle Strength, and Cognitive Function in Patients Diagnosed With Schizophrenia
Status: Completed | Type: Observational
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, İsmail Koç, Assistant Prof, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: Ismail KKoc
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-08

CONDITIONS: Schizophrenia Disorder
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with schizophrenia: patients with schizophrenia

SUMMARY:
Schizophrenia is a serious mental health condition that affects individuals' thinking, perception, emotional responses, and behavior.

Balance in schizophrenia patients is often related to motor skills, coordination, and postural control.

Schizophrenia can cause functional changes in certain areas of the brain. These changes can affect motor functions.

Balance loss in schizophrenia patients can cause difficulties in daily living activities, increased risk of falls, and a decrease in overall quality of life. Therefore, the aim of this study is to evaluate physical activity, balance, muscle strength, and cognitive function in patients diagnosed with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a serious mental health condition that affects individuals' thinking, perception, emotional responses, and behavior. Treatment for schizophrenia typically involves approaches such as medication and psychotherapy. Balance in schizophrenia patients is often related to motor skills, coordination, and postural control. Although schizophrenia is a mental health disorder, it can also affect patients' physical balance and motor function. Antipsychotic medications, which are frequently used in the treatment of schizophrenia, can have an effect on patients' motor skills. These medications can negatively affect balance in some patients.

Schizophrenia can cause functional changes in certain areas of the brain. These changes can affect motor functions. Hallucinations, which are commonly seen in patients with schizophrenia, can interfere with visual, auditory, or tactile perception, preventing the person from accurately perceiving their surroundings. This can negatively affect physical balance, as the person may not be able to accurately assess dangers in their surroundings or may misperceive their location or distances. Balance loss in schizophrenia patients can cause difficulties in daily living activities, increased risk of falls, and a decrease in overall quality of life. Therefore, the aim of this study is to evaluate physical activity, balance, muscle strength, and cognitive function in patients diagnosed with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia by a psychiatrist according to DSM-V
* Unchanged medication treatment for the last 2 months
* Being over 18 years of age
* Individuals must be able to understand and speak Turkish
* Individuals must be able to read and write

Exclusion Criteria:

* Uncontrolled hypertension
* Surgery within the last 2 months
* Orthopedic surgery on the lower extremities
* Cardio-respiratory failure that prevents walking

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with Schizophrenia
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2025-08-19 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale | 2 weeks
  This is a 30-item, 7-point semi-structured interview scale. Of the 30 psychiatric parameters, seven belong to the positive symptoms subscale, seven to the negative symptoms subscale, and 16 to the general psychopathology subscale. The Turkish reliability and validity study of the scale was conducted by Kostakoğlu et al.
Mini Mental State Examination | 2 weeks
  The standardized version of the MMSE (Mini Mental State Examination) developed by Folstein et al. (1975) was adapted by Molloy and Standish (1997). The MMSE allows for cognitive assessment in a short period of time. In this regard, the MMSE is a short, easy-to-administer, and standardized test used to assess global cognitive level. The test is widely used to evaluate the cognitive status of elderly individuals. A validity and reliability study in the Turkish population was conducted by Güngen and colleagues (2002). In their study, Güngen and colleagues (2002) determined that the 23/24 cutoff value of the Standardized Mini Mental Test (SMMT) had a sensitivity of 0.91, a specificity of 0.95, an inter-rater reliability of r:0.99, and a kappa value of 0.92. As a result, it was determined that the Standardized Mini Mental Test is valid and reliable in the Turkish population.
Handgrip Strength | 2 weeks
  The Jamar hand dynamometer, recommended by the American Hand Therapy Association (AETD) and widely accepted as the gold standard due to its high validity and reliability in numerous studies, will be used to measure hand grip strength. Hand grip strength will be measured in the standard position recommended by the ATA: sitting position, shoulders in adduction and neutral rotation, elbow at 90° flexion, forearm in mid-rotation and supported, wrist in neutral position. In the test procedure, three measurements will be taken for handgrip strength, with one-minute intervals between each measurement, and the averages will be recorded.
Berg Balance Scale | 2 weeks
  Berg Balance Scale The scale, consisting of a total of 14 items, assesses patients' balance skills. Each item is scored on a scale of 0-4. 0 = unable to perform, 4 = normal performance. The maximum score is 56, and a high score indicates better balance skills. The physical therapist administers the test by providing the necessary instructions to the patient in a manner they can understand after the patient has rested. The choice of which foot to use in certain items should be left to the patient. The materials required for the test (stopwatch, measuring tape, chair, step, slippers) should be prepared before beginning the assessment.
30-Second Sit-to-Stand Test | 2 weeks
  The individual will be positioned in the center of the chair with their back straight, feet flat on the ground, and arms crossed in front of their chest (right hand on left shoulder, left hand on right shoulder). In this position, the test will begin with the command "start," and the subject will perform as many full stand-ups as possible within 30 seconds. The number of full stand-ups performed within 30 seconds will constitute the subject's score. To ensure the test is performed safely, the back of the chair will be secured against a wall or a sturdy surface. Each participant will be shown how to perform the test, and after ensuring that they understand how to perform the test by having them attempt it 2-3 times, the test will begin.
International Physical Activity Questionnaire (IPAQ): | 2 weeks
  Used to assess an individual's physical activity level over the past 7 days. The International Physical Activity Questionnaire (IPAQ) consists of 4 questionnaires. There are long (5 independently asked activity areas) and short (4 general items) versions. The short version consists of questions about the time spent walking and engaging in moderate to vigorous and strenuous activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Dr Lütfi Kırdar City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No